CLINICAL TRIAL: NCT00005355
Title: Gender Differences in Familial Risk
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4241; R01HL048148 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

SUMMARY:
To develop, test, and apply comprehensive mathematical models for the interaction of genetic and environmental effect on cardiovascular risk with gender differences.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

Models were developed which allowed for sex difference in the expression of autosomal polygenes, differences in the impact of the paternal and maternal environment on male and female offspring, and for the complex consequences of assortative mating on the correlations among loci and between genes and environment. Computer simulations were used to decide which kinds of gender-dependent effects could be resolved with particular constellations of relatives, and to address problems of power and bias resulting from errors of model-specification. The methods developed were applied to data from extensive data already gathered from twins and their relatives to determine the importance of sex differences in genetic and environmental causes of variation in measured aspects of cardiovascular risk including weight, body-mass index, family history of CV disease, smoking, alcohol consumption, exercise, diet, psychosocial variables and lifestyle.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1993-02; Study Completion 1996-01

REFERENCES:
- [Background] Loos R, Thomis M, Maes HH, Beunen G, Claessens AL, Derom C, Legius E, Derom R, Vlietinck R. Gender-specific regional changes in genetic structure of muscularity in early adolescence. J Appl Physiol (1985). 1997 Jun;82(6):1802-10. doi: 10.1152/jappl.1997.82.6.1802. PMID 9173944
- [Background] Thomis MA, Van Leemputte M, Maes HH, Blimkie CJ, Claessens AL, Marchal G, Willems E, Vlietinck RF, Beunen GP. Multivariate genetic analysis of maximal isometric muscle force at different elbow angles. J Appl Physiol (1985). 1997 Mar;82(3):959-67. doi: 10.1152/jappl.1997.82.3.959. PMID 9074988
- [Background] Maes HH, Beunen GP, Vlietinck RF, Neale MC, Thomis M, Vanden Eynde B, Lysens R, Simons J, Derom C, Derom R. Inheritance of physical fitness in 10-yr-old twins and their parents. Med Sci Sports Exerc. 1996 Dec;28(12):1479-91. doi: 10.1097/00005768-199612000-00007. PMID 8970142
- [Background] Eaves LJ, Neale MC, Maes H. Multivariate multipoint linkage analysis of quantitative trait loci. Behav Genet. 1996 Sep;26(5):519-25. doi: 10.1007/BF02359757. PMID 8917951
- [Background] Meyer JM, Han J, Singh R, Moxley G. Sex influences on the penetrance of HLA shared-epitope genotypes for rheumatoid arthritis. Am J Hum Genet. 1996 Feb;58(2):371-83. PMID 8571964
- [Background] Neale MC, Eaves LJ, Kendler KS. The power of the classical twin study to resolve variation in threshold traits. Behav Genet. 1994 May;24(3):239-58. doi: 10.1007/BF01067191. PMID 7945154
- [Background] Neale MC, Walters EE, Eaves LJ, Maes HH, Kendler KS. Multivariate genetic analysis of twin-family data on fears: Mx models. Behav Genet. 1994 Mar;24(2):119-39. doi: 10.1007/BF01067816. PMID 8024529
- [Background] Eaves LJ. Effect of genetic architecture on the power of human linkage studies to resolve the contribution of quantitative trait loci. Heredity (Edinb). 1994 Feb;72 ( Pt 2):175-92. doi: 10.1038/hdy.1994.25. PMID 8150657